CLINICAL TRIAL: NCT04297891
Title: Phenotypes, Biomarkers and Pathophysiology in Spastic Ataxias
Acronym: SPAX-PBP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Rebecca Schule (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other); German Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Dr. Rebecca Schule, Principal Investigator, Leading Consultant, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Other Study IDs: SPAX-PBP; 441409627 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2020-02-27; First posted 2020-03-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Spastic Ataxia
Keywords: Spastic Ataxia; Biomarker; Genetic etiology; Molecular mechanisms; Natural History Study
MeSH Terms: conditions — Spastic Ataxia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — optional biosample collection including blood (DNA, serum, plasma, RNA, PBMC), urine, CSF, skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARSACS: Participants with genetically confirmed ARSACS (ORPHA:98) will be recruited. Target sample size for the ARSACS cohort is 120.
  Interventions: Other: Clinical rating scale to measure Ataxia disease severity and progression; Other: Clinical rating scale to measure spastic paraplegia disease severity and progression; Other: Disease-specific severity index for adults with autosomal recessive spastic ataxia of Charlevoix-Saguenay (ARSACS); Diagnostic Test: Next-Gen Sequencing (NGS)
- SPG7: Participants with genetically confirmed SPG7 (ORPHA:99013) will be recruited. Target sample size for the SPG7 cohort is 72.
  Interventions: Other: Clinical rating scale to measure Ataxia disease severity and progression; Other: Clinical rating scale to measure spastic paraplegia disease severity and progression; Other: Disease-specific severity index for adults with autosomal recessive spastic ataxia of Charlevoix-Saguenay (ARSACS); Diagnostic Test: Next-Gen Sequencing (NGS)
- Unrelated healthy control: Unrelated healthy controls Healthy controls may undergo the same study procedures as the ARSACS and SPG7 cohort. Target sample size for the control cohort is 50.
  Interventions: Other: Clinical rating scale to measure Ataxia disease severity and progression; Other: Clinical rating scale to measure spastic paraplegia disease severity and progression; Other: Disease-specific severity index for adults with autosomal recessive spastic ataxia of Charlevoix-Saguenay (ARSACS); Diagnostic Test: Next-Gen Sequencing (NGS)

INTERVENTIONS:
Other: Clinical rating scale to measure Ataxia disease severity and progression — SARA is a clinical scale developed by Schmitz-Hübsch et al which assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
  Other Names: Scale for the Assessment and rating of Ataxia (SARA)
Other: Clinical rating scale to measure spastic paraplegia disease severity and progression — A 13-item scale to rate functional impairment occurring in pure forms of spastic paraplegia (SP). Additional symptoms constituting a complicated form of SP are recorded in an inventory.
  Other Names: Spastic Paraplegia Rating Scale (SPRS)
Other: Disease-specific severity index for adults with autosomal recessive spastic ataxia of Charlevoix-Saguenay (ARSACS) — The DSI-ARSACS is a valid measure of disease severity for the adult ARSACS population that is able to distinguish between patients with different clinical profiles.
  It considers the 3 components (pyramidal, cerebellar, neuropathic) of the disease, and documents its content validity, internal consistency, and construct validity.
  Other Names: DSI-ARSACS
Diagnostic Test: Next-Gen Sequencing (NGS) — Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Spastic Ataxias (SPAX) and related disorders in a prospective multicenter natural history study, identify digital, imaging and molecular biomarkers that can assist in diagnosis and therapy development and study the genetic etiology and molecular mechanisms of these diseases.

DETAILED DESCRIPTION:
The investigators will perform a registry-based standardized prospective Natural History Study (NHS) in SPAX and related disorders. Participants will be seen annually. At study visits a standardized clinical examination will be performed including application of clinical rating scales (selection of rating scales may vary depending on the individual phenotype and specific genotype); data will be entered into a clinical database (HSP Registry; https://www.hsp-registry.net and ARCA Registry; www.ARCA-registry.org). At all study visits, patients will be asked to donate biosamples; biomaterial collection is optional and participants can elect to participate in sampling of blood, urine, CSF, and/or a skin biopsy.

Optionally, additional examinations may be performed including imaging, quantitative movement analysis, neuropsychological examinations, analysis of patient or observer reported outcomes and OMICS analysis to characterize molecular biomarkers.

In participants without a genetic diagnosis, next generation sequencing may be performed.

Thus this study will establish a model of disease progression and mechanistic evolution in SPAX, which will allow to track and understand selective as well as overlapping dysfunction of the cerebellum and corticospinal tract. In a transatlantic natural history study we will longitudinally validate clinician- and patient-reported, digital and molecular outcomes. In addition, we will improve on existing and develop new outcome parameters that show superior sensitivity to change. These include a novel clinical SPAX composite score, a smartphone mHealth toolbox combining remote assessment of daily living by wearable sensors with app-based patient-entered outcomes (SPAX.app), and multimodal MRI radiomics with an innovative machine learning approach for multisite MRI analysis, including in particular the infratentorial space. Longitudinal validation of targeted fluid biomarker candidates will aslo be an important part.

ELIGIBILITY:
Inclusion Criteria:

* ARSACS cohort: genetic diagnosis of ARSACS and clinically manifest disease
* SPG7 cohort: genetic diagnosis of SPG7 and clinically manifest disease
* Unrelated healthy controls: no signs or history of neurological or psychiatric disease

AND

* written informed consent provided

AND

* Participants are willing and able to comply with study procedures

Exclusion Criteria:

* Missing informed consent
* For controls: evidence of a neurodegenerative disease or movement disorders; inability to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Probands with clinically manifest and genetically confirmed spastic ataxia (genetic subtypes: ARSACS, SPG7) will be enrolled in this study. Additionally, healthy unrelated controls will be enrolled; these are necessary to contrast unspecific, gender- or age-related findings to disease specific findings.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change of Scale for the Assessment and Rating of Ataxia (SARA) from baseline to 2-year follow-up | 24 months
  Severity of the ataxia component of the disease will be assessed by application of the Scale for the Assessment and Rating of Ataxia (SARA). The total score is calculated as the sum of al items, yielding a total score between 0 and 38. Hereby, higher SARA scores indicate more severe disease.
Change of Spastic Paraplegia Rating Scale (SPRS) from baseline to 2-year follow-up | 24 months
  Severity of the spasticity component of the disease will be assessed by application of the Spastic Paraplegia Rating Scale. The total score is calculated as the sum of al items, yielding a total score between 0 and 52. Hereby, higher SPRS scores indicate more severe disease.

SECONDARY OUTCOMES:
Change of Disease severity index - Autosomal recessive spastic ataxia of Charlevoix-Saguenay(DSI-ARSACS) from baseline to 2-year follow-up | 24 months
  The DSI-ARSACS is a clinical rating scale consisting of 8 items reflecting the 3 main components of the disease (pyramidal, cerebellar, and neuropath systems) specifically developed to measure disease progression in ARSACs. The DSI-ARSACS total score can range from 0 to 38. Hereby, higher DSI-ARSACS scores indicate more severe disease.

OTHER OUTCOMES:
Change of the Patient-Reported Outcomes Measurement Information System (PROMIS) short form "physical function" 12a from baseline to 2-year follow-up | 24 months
  Self-report questionnaire comprising 12 questions. All PROMIS scores are standardized (item-level calibration) and expressed as T-scores with a population mean of 50 and a Standard Deviation (SD) of 10. Higher T-scores hereby indicate a higher physical function level.
Change of the Patient-Reported Outcomes Measurement Information System (PROMIS) short form "social roles and activities" 8a from baseline to 2-year follow-up | 24 months
  Self-report questionnaire comprising 8 questions. All PROMIS scores are standardized (item-level calibration) and expressed as T-scores with a population mean of 50 and a Standard Deviation (SD) of 10. Higher T-scores hereby indicate a higher degree of social participation.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schüle, PD Dr., Principal Investigator — University Hospital Tübingen; Matthis Synofzik, Prof., Dr., Principal Investigator — University Hospital Tübingen
Locations (9):
- Canada (2):
  - Montreal Neurological Institute of McGill University, Department of Neurology and Neurosurgery and Human Genetics, Montreal, Quebec
  - Université de Sherbrooke, Saguenay, Quebec
- Département d'information médicale (DIM); Département de Biostatistique, Santn 3emé Publique et Information Médicale (BIOSPIM)- Bâtiment Mazarie étage; Hôpitaux Universitaires Pitié Salpêtrière, Paris, France
- Germany (2):
  - Center for Neurology & Hertie-Institute for Clinical Brain Research, Dept. for Neurodegenerative Diseases, Tübingen, Baden-Wurttemberg
  - University Hospital Essen (AöR), Essen
- IRCCS Fondazione Stella Maris, Pisa, Italy
- Radboud University Medical Center; Department of Neurology & Donders Institute for Brain, Cognition, and Behaviour, Nijmegen, Netherlands
- Koç Univ. Hospital, KUTTAMNDAL, Istanbul, Turkey (Türkiye)
- Department of Clinical Neurosciences, University of Cambridge; John Van Geest Cambridge Centre for Brain Repair, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamdan A, Traschutz A, Beichert L, Chen X, Gagnon C, van de Warrenburg BP, Santorelli FM, Basak N, Coarelli G, Horvath R, Klebe S; PROSPAX consortium; EVIDENCE-RND consortium; Schule R, Hooker AC, Synofzik M, Karlsson MO. Integrated Modeling of Digital-Motor and Clinician-Reported Outcomes Using Item Response Theory: Towards Powerful Trials for Rare Neurological Diseases. CPT Pharmacometrics Syst Pharmacol. 2025 Nov;14(11):1857-1868. doi: 10.1002/psp4.70081. Epub 2025 Jul 21. PMID 40685914
- See also: Website of the HSP Registry — http://treathsp.net
- See also: Website of the ARCA Registry — http://arca-registry.org